CLINICAL TRIAL: NCT06075251
Title: Stepped-Care Online Parent Support Following Congenital Heart Disease: A Randomized Control Trial
Brief Title: Online Support 4 CHD Kids & Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Tricia Williams, Associate Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000080752
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: This study is a single-site, two-arm randomized clinical trial. Families will be randomized to receive care as usual or active I-InTERACT-North stepped-care treatment.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors responsible for coding the primary outcome will be masked to condition. Due to the nature of the intervention (behavioural program), participants and care providers cannot be masked to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I-InTERACT-North (Experimental): Virtual stepped-care positive parenting program.
  Interventions: Behavioral: I-InTERACT-North
- Care as Usual (No Intervention): The CAU group will receive no direct parent treatment other than clinical care provided in cardiac follow-up (i.e., child assessment and consultation), which will be documented at each follow up. At end of trial, participants randomized to CAU will have the option to participate in I-InTERACT-North.

INTERVENTIONS:
Behavioral: I-InTERACT-North — I-InTERACT-North is a virtual stepped-care positive parenting program. It comprises online psychoeducational modules as well as live therapy and coaching sessions. The program lasts anywhere from 1 to 16 weeks depending on parents' progress.
  Arms: I-InTERACT-North

SUMMARY:
This study will evaluate a virtual mental health parenting stepped-care intervention (I-InTERACT-North) to determine if the program works to improve positive parenting skills and child behaviour among families with children born with Congenital Heart Disease (CHD). Recruitment will target children ages 3-9 years old from SickKids. We will also evaluate the acceptability and feasibility of the program among children and families to inform future delivery and multi-site trials. Results will evaluate whether I-InTERACT-North can improve parenting and child behaviour in these families and inform future best clinical practices for this population.

DETAILED DESCRIPTION:
The proposed Hybrid Type 1 study is a single-site, two-arm single blinded randomized clinical trial (RCT) designed to simultaneously assess: 1) efficacy of the stepped care I-InTERACT-North program in improving positive parenting skills and child behaviour among families of children with Congenital Heart Disease (CHD) and 2) feasibility and acceptability outcomes (i.e., adherence, fidelity, costs and acceptability). Our primary aim is to determine the efficacy of the I-InTERACT-North stepped-care program compared to care as usual in improving positive parenting skills (primary outcome) and reducing child emotional and behavioural problems (co-primary outcome) among CHD children. Our secondary aim is to examine feasibility and acceptability of the stepped-care program among key stakeholders (parents, therapists, medical providers). Our exploratory aim is to examine the association between neonatal white matter injury severity on treatment and implementation outcomes.

The study population will be parents of children currently ages 3 to 9 with histories of Congenital Heart Disease and are part of existing research cohorts (Cardiovascular Physiology and Brain Development in Neonates with Congenital Heart Disease; Pediatric Cardiac and Neurological Registry at SickKids) and have consented to be contacted for future studies.

I-InTERACT-North is an evidenced-based virtual parenting skills training program, which emphasizes building a warm, responsive relationship between parent and child and establishing guidelines for consistent behaviour management. It also provides education on the effects of medical conditions on children's learning and behaviour. The stepped-care program provides three steps that sequentially increase therapy content and degree of therapist involvement, (1) Psychoeducation-Podcast, (2) Intro to Positive Parenting (2 coaching sessions), and (3) Full Program (5 coaching sessions). Coaching sessions are offered via videoconference weekly or biweekly based on parent availability.

A care as usual (CAU) was chosen as the optimal comparator given its alignment with the primary research question, and consistent with prior studies of the program. The CAU group will receive no direct parent treatment other than clinical care provided in cardiac follow-up (i.e., child assessment and consultation), which will be documented at each follow up. At end of trial, the CAU will be offered the program.

All consenting participants will complete baseline questionnaires. Following consent and completion of baseline measures (therefore hidden allocation), participants will be randomized by a research coordinator independent of our intervention team. Randomization will be balanced by 1) child sex assigned at birth, and 2) baseline child behaviour concern intensity (based on median split grouping; pilot study ECBI median t-score =60.00). All participants will complete follow-up questionnaires at 3 months, 6 months, and 12 months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child aged 3 to 9 years with history of congenital heart disease
* Parent of a patient at The Hospital for Sick Children (SickKids)
* Resident of Ontario, Canada

Exclusion Criteria:

* Significant major medical issues requiring ongoing inpatient care (e.g., children participating in significant surgical or inpatient treatment)
* Current participation in an equivalent family/parent therapy program (e.g., Incredible Years Parenting Program (IYPP), Positive Parenting Program (Triple P))
* Previous participation in an I-InTERACT-North pilot study

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 382 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive Parenting Skills | Baseline, 3 months, 6 months, and 12 months
  The primary proximal outcome will be positive parenting skills assessed through blinded (to allocation and follow up interval) coding of recorded parent-child interactions, using the Dyadic Parent-Child Interaction Coding System (DPICS). The DPICS will be used to rate positive parenting behaviors (e.g. praise, responsiveness, and enthusiasm). The DPICS is analyzed by independent blinded coders (to condition and time) observe and code parent-child interactions (5 minutes) for positive parenting behaviours (e.g., praise, responsiveness and enthusiasm).
Child Behaviour | Baseline, 3 months, 6 months, and 12 months
  The Eyberg Child Behavior Inventory (ECBI), is a parent rated 36-item checklist of concerns (e.g., noncompliance, emotional regulation).

SECONDARY OUTCOMES:
Quality of Life | Baseline, 3 months, 6 months, and 12 months
  Parent reports of their child and family's Quality of Life (QoL) will be evaluated with EuroQol 5 Dimensions 5 Levels questionnaire (EQ5D-5L), previously used in the context of parent stress with favourable psychometric properties, and items related to child internalizing symptoms, i.e., anxiety/ depression, self-care and daily activities.
Parent Mental Health | Baseline, 3 months, 6 months, and 12 months
  The Depression Anxiety and Stress Scale Short Form (DASS-21) is a self-report measure of mental health and includes three subscales (depression, anxiety, and stress). Parents rate a series of 21 statements describing depression, anxiety, and stress on a scale of 0 to 3. Higher scores on the DASS indicate greater mental health concerns.
Service Utilisation | Baseline, 3 months, 6 months, and 12 months
  The Client Services Receipt Inventory (CSRI) includes questions for parents regarding the child and family's use of mental health, community rehabilitation, neuropsychology, and educational psychology services as well as paid and unpaid caregiver time and time off work.

CONTACTS AND LOCATIONS:
Overall Officials: Tricia S Williams, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taylor M, Bondi BC, Andrade BF, Au-Young SH, Chau V, Danguecan A, Desire N, Guo T, Ostojic-Aitkens D, Wade S, Miller S, Williams TS. Stepped-Care Web-Based Parent Support Following Congenital Heart Disease: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Oct 4;13:e64216. doi: 10.2196/64216. PMID 39365658